CLINICAL TRIAL: NCT01750411
Title: The Severe Asthma Research Program at Wake Forest University - Longitudinal Phenomics and Genetics of Severe Asthma.
Brief Title: Severe Asthma Research Program - Wake Forest University
Acronym: SARP3
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: IRB00021507; 1U10HL109164-01 (NIH)
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-02

CONDITIONS: Asthma; Severe Persistent Asthma
Keywords: Severe Asthma; SARP
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood: CBC/Diff, Total IgE, Serum, Plasma, DNA, RNA Urine EBC Sputum: Supernatant, Cell Pellet Bronch: BAl, Bronchial Brushings, Bronchial Biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asthma: Severe Asthma Not severe Asthma

SUMMARY:
The mission of SARP is to improve the understanding of severe asthma through the integrated study of the effect of genetics on the clinical and biological features of asthma and to investigate how these change over time. The ultimate goal of these efforts is to promote better treatments for severe asthma.

DETAILED DESCRIPTION:
The mission of the SARP is to improve the understanding of severe asthma to develop better treatments. The SARP will gain a better understanding of asthma and its endotypes, in children and adults, by defining the disease at the molecular and cellular levels in the context of the temporal phenotypic expression of the disease. To this end, the SARP investigators will utilize both mechanistic and evoked phenotype approaches to: 1) characterize developmental molecular, cellular and physiologic phenotypes in children and adults with mild to severe asthma, and 2) to further elucidate the evolving pathobiology and pathogenesis of severe asthma and its sub-phenotypes and 3) compare these features over time. This approach involves a shared longitudinal protocol conducted across all participating centers which includes common information on all SARP participants. Additionally, SARP investigators have each identified mechanistic research questions to be included in the shared longitudinal protocol. At Wake Forest University investigators are specifically interested in genetic influences on disease severity and the use of statistical modeling techniques to better understand disease phenotypes. Together, these longitudinal and mechanistic approaches will enable prediction of phenotype stability/fluctuation and pharmacologic responses and identification of novel, disease-modifying targets for treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Physician diagnosis of asthma,
2. Age 6 years and older
3. Evidence of historical reversibility, including either:

   * FEV1 bronchodilator reversibility ≥ 12%, or
   * Airway hyperresponsiveness reflected by methacholine PC20≤16 mg/mL.

Exclusion Criteria:

1. No primary medical caregiver
2. Pregnancy (only if undergoing methacholine challenge or bronchoscopy)
3. Current smoking
4. Smoking history > 10 pack years if ≥ 30 years of age or smoking history >5 pack years if < 30 years of age (Note: If a subject has a smoking history, no smoking within the past year)
5. Other chronic pulmonary disorders associated with asthma-like symptoms, including (but not limited to) cystic fibrosis, chronic obstructive pulmonary disease, chronic bronchitis, vocal cord dysfunction that is the sole cause of asthma symptoms, severe scoliosis or chest wall deformities that affect lung function, or congenital disorders of the lungs or airways
6. History of premature birth before 35 weeks gestation
7. Planning to relocate from the clinical center area before study completion

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target recruitment goal for each center is 75% adults (age 18 and older) and 25% children age 6-17 years. Within the pediatric age group, an attempt will be made to enroll equal numbers of children 6-11 and 12-17 years of age. Similarly, an attempt will be made to enroll at least 50% females and 30% minorities.
  Given the mission of SARP, a diverse sample of subjects with asthma is needed to gain better understanding of asthma and its endotypes. Because there are a number of respiratory disorders that may be confused with asthma or confound asthma assessment, SARP enrollees must meet the all following eligibility criteria as outlined below:
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2012-12; Primary Completion 2020-02-18 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Change in pulmonary function over time | 36 months
  Pulmonary function test results include forced expiratory volume in one second (FEV1) and forced vital capacity (FVC).

SECONDARY OUTCOMES:
Frequency of severe asthma exacerbations | 36 months
  Frequency of severe asthma exacerbations
  * Utilization of hospital based care (Emergency Department, Hospitalization, ICU)
  * Need for supplemental oral corticosteroids

CONTACTS AND LOCATIONS:
Overall Officials: Eugene R Bleecker, MD, Principal Investigator — University of Arizona Department of Medicine; Deborah A Meyers, PhD, Principal Investigator — University of Arizona Department of Medicine; Wendy C Moore, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Huang BK, Elicker BM, Henry TS, Kallianos KG, Hahn LD, Tang M, Heng F, McCulloch CE, Bhakta NR, Majumdar S, Choi J, Denlinger LC, Fain SB, Hastie AT, Hoffman EA, Israel E, Jarjour NN, Levy BD, Mauger DT, Sumino K, Wenzel SE, Castro M, Woodruff PG, Fahy JV, Sarp FTNSARP. Persistent mucus plugs in proximal airways are consequential for airflow limitation in asthma. JCI Insight. 2024 Feb 8;9(3):e174124. doi: 10.1172/jci.insight.174124. PMID 38127464
- [Derived] Dunican EM, Elicker BM, Gierada DS, Nagle SK, Schiebler ML, Newell JD, Raymond WW, Lachowicz-Scroggins ME, Di Maio S, Hoffman EA, Castro M, Fain SB, Jarjour NN, Israel E, Levy BD, Erzurum SC, Wenzel SE, Meyers DA, Bleecker ER, Phillips BR, Mauger DT, Gordon ED, Woodruff PG, Peters MC, Fahy JV; National Heart Lung and Blood Institute (NHLBI) Severe Asthma Research Program (SARP). Mucus plugs in patients with asthma linked to eosinophilia and airflow obstruction. J Clin Invest. 2018 Mar 1;128(3):997-1009. doi: 10.1172/JCI95693. Epub 2018 Feb 5. PMID 29400693
- See also: Severe Asthma Research Program Public Website — http://severeasthma.org/

DOCUMENTS (1):
  • Informed Consent Form (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT01750411/ICF_000.pdf